CLINICAL TRIAL: NCT00782873
Title: Balanced Propofol Sedation During Upper Endoscopy in Morbidly Obese Patients: Assessment of Cardiopulmonary Parameters
Brief Title: Balanced Propofol Sedation During Upper Endoscopy in Morbidly Obese Patients
Status: Completed | Type: Observational
Sponsor: Research Associates of New York, LLP (Other)
Responsible Party: Lawrence B. Cohen, MD, Research Associates Of New York
Other Study IDs: 424-02-08
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Obesity
Keywords: propofol; sedation; safety; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- obese subjects: BMI > 35

SUMMARY:
The purpose of this study is to evaluate the safety of propofol-based, gastroenterologist-administered sedation in severely obese patients (BMI≥35) undergoing upper endoscopy.

The investigators aim to test the hypothesis that it is safe to use balanced-propofol, gastroenterologist-administered sedation in obese patients.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety of propofol-based, gastroenterologist-administered sedation in severely obese patients (BMI≥35) undergoing upper endoscopy. We will use changes in pulmonary and hemodynamic parameters as the primary safety measure in this study. We will compare these results in 30 non-obese patients and in 30 obese patients.

The term balanced propofol sedation refers to using a low dose of propofol in combination with small amounts of an opioid and midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an endoscopic esophagostroduodenoscopy (EGD)
* Capable of providing written informed consent and willing and able to comply with all procedures of the study
* Adults between the ages of 18 and 85 inclusive (and of legal age to consent)
* ASA score of I, II, or III

Exclusion Criteria:

* Severe acute illness that is not resolved or stabilized prior to enrollment. Study entry will be based on the investigator's judgment
* Need for sleep or narcotic analgesic medication on a continuous basis during the proceeding 6 months
* Pregnancy
* A history of drug addiction or alcohol abuse within the past 12 months. Alcohol can be consumed in moderation. The consumption of alcohol should be within the routine pattern for the individual before the study.
* A history of seizure disorder.
* Allergy to propofol, soy beans, or eggs.
* Prior history of difficult intubation.
* Prior history of severe complications during conscious sedation. Study entry will be based on the investigator's judgment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research subjects will be selected from a private practice.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
A change in mean arterial pressure (MAP) of 20% or more from baseline | during upper endoscopy

SECONDARY OUTCOMES:
Episodes of bradycardia - pulse less than 50 | during upper endoscopy
ECG changes consistent with myocardial ischemia | during upper endoscopy
Decrease in respiratory rate - change of 20% or more from baseline | during upper endoscopy
Assess the dose of propofol, midazolam, and fentanyl necessary to achieve adequate sedation during upper endoscopy and compare the dose requirements of the obese and non-obese patient cohorts. | after all patients completed
Compare the level of sedation between the obese and non-obese cohorts | after all patients completed
compare patient satisfaction with endoscopic sedation in obese and non-obese cohorts | after all patients completed
Compare time to sedation in the obese and non-obese cohorts | after all patients completed
Oxygen desaturation | during upper endoscopy
Apneic episodes | during upper endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence B Cohen, MD, Principal Investigator — Research Associates of New York
Locations (1):
- Research Associates of New York, New York, New York, United States